CLINICAL TRIAL: NCT05854940
Title: Multicenter, Prospective Clinical Study of the Serum Raman Spectroscopy Intelligent System for the Diagnosis of Prostate Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Changhai Hospital (Other); Ruijin Hospital (Other); Tongji Hospital (Other); Peking University People's Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: LY2023-026-B
Record Dates: First submitted 2023-04-26; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Raman spectroscopy; Early diagnosis; artificial intelligence
MeSH Terms: conditions — Prostatic Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Eligible participants for early diagnosis of prostate cancer: According to the 2014 edition of China Prostate Cancer Diagnosis and Treatment Guidelines, patients need to undergo prostate biopsy
  Interventions: Diagnostic Test: Serum Raman spectroscopy intelligent diagnostic system

INTERVENTIONS:
Diagnostic Test: Serum Raman spectroscopy intelligent diagnostic system — Intelligent diagnostic system based on Raman spectrum of serum

SUMMARY:
At present, the most commonly used clinical screening tool is based on prostate-specific antigen (PSA) examination. Because PSA is a tissue-specific rather than a tumor-specific marker, it has low specificity and sensitivity for prostate cancer. Although these PSA-related diagnostic models (PHI, 4Kscore) have been proved to improve the sensitivity and specificity of the early diagnosis of prostate cancer, they still do not meet the requirements of accurate diagnosis. Therefore, it is extremely important to develop a diagnosis tool with higher specificity, sensitivity and accuracy in the current prostate tumor screening strategy.

Raman spectroscopy (Raman Spectrum, RS) as a non-invasive and high specificity of material molecular detection technology, can be obtained in the molecular level, thus sensitive to detect biological samples tumor metabolism related proteins, nucleic acids, lipids and sugar composition of bio-molecules changes. As scientists pointed out in a literature in "chemical society reviews"in 2020, although SERS technology has shown good diagnostic efficacy in lots of preclinical studies in multiple tumors, it is limited to a generally small sample size and lacks external validation. There for, a clinical study of Raman spectra for tumor diagnosis is needed, which meets the following requirements: 1.An objective, fast and practical application of Raman spectral data processing is needed and deep learning method may be the best classification method; 2. It requires multicenter and large clinical samples to train deep learning diagnostic model, and verify its true efficacy through external data of prospective study.

In our preliminary study,we have collected Raman spectra data from a large cohort of 2899 patients and constructed Raman intelligent diagnostic system based on CNN model. The intelligent diagnostic system achieved accuracy of 83%. In order to obtain the highest level of clinical evidence and truly realize clinical transformation, this prospective, multi-center clinical study is designed to verify the intelligent diagnostic system for early diagnosis of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with suspected prostate cancer and meet the Chinese Guidelines for Prostate Cancer (2014 edition)
2. PSA≤20;
3. The ECGO score was 0-1, and the cardiopulmonary function tolerated prostate biopsy;
4. After being fully informed of the purpose and possible risks of the study, the patient agrees to participate in the trial and signed the "Informed Consent for the use of clinical samples".

Exclusion criteria:

1. Previous history of other cancer;
2. Metabolic disorders caused by chronic renal failure or metabolic diseases, obviously abnormal blood sugar, blood lipid and plasma protein;
3. Previously taking 5- α reductase inhibitor drug;
4. History of acute prostatitis or minimally invasive surgery inside the prostate cavity for 3 months prior to puncture;
5. History of multiple blood transfusion;
6. Failure to cooperate with or refuse to participate in the clinical trial later.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected prostate cancer and meet the Chinese Guidelines for Prostate Cancer (2014 edition); including:
  1. Digital rectal examination found prostate nodules, any PSA.
  2. B ultrasound, CT, MRI found abnormal signals, any PSA.
  3. PSA> 10 ng/ml, any f / t PSA and PSAD values.
  4. PSA 4 ~ 10 ng/ml, abnormal f / t PSA value or abnormal PSD value.
Sampling Method: Non-Probability Sample
Enrollment: 490 (Estimated)
Dates: Start 2023-06-10 (Estimated); Primary Completion 2023-06-10 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The accuracy of the Serum Raman Spectroscopy Intelligent System | 2023.6
  According to the final pathology results of prostate biopsy, count the accuracy of Serum Raman Spectroscopy Intelligent System for prostate cancer diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- RenJi hospital, school of Medicine, Shanghai Jiao Tong University, Shanghai, China